CLINICAL TRIAL: NCT06789926
Title: The Impact of Multimedia Psychological Support Platform and Acceptance and Commitment Therapy Workshops on the Mental and Physical State of Oncology Nurses
Brief Title: The Impact of Multimedia Psychological Support Platform and Acceptance and Commitment Therapy Workshops of Oncology Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202411009RIND
Record Dates: First submitted 2024-12-05; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Oncology Nurse; Psychological Support; Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Other): After attending a 4-hour ACT workshop, participants will utilize the remaining course time to independently access the LINE platform. The platform will feature pre-recorded guided audio files for relaxation, emotional videos, and psychological cards.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — Attending a 4-hour ACT workshop, and after attending participants will utilize the remaining course time to independently access the LINE platform. The platform will feature pre-recorded guided audio files for relaxation, emotional videos, and psychological cards.

SUMMARY:
Based on the high levels of emotional distress, burnout, and turnover intentions among clinical oncology nursing staff, this study will provide a multimedia "Mind-Body Support" Line platform and ACT workshop courses as intervention measures for oncology nursing staff. The study aims to explore the effectiveness of these interventions in alleviating their psychological and physical distress, utilizing both qualitative and quantitative research methods to achieve the research objectives.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as an oncology nurse in a clinical setting

Exclusion Criteria:

* "Unwilling or unable to participate in the full training course"

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological flexibility | Measurements will be taken before the workshop intervention, immediately after the workshop intervention, and one month later.
  We utilized the Work-related Acceptance and Action Questionnaire (WAAQ) as the primary outcome measure. This scale assesses psychological resilience in the workplace and comprises 7 items, each rated on a 7-point Likert scale. A score of 1 indicates that the described situation never applies, while a score of 7 indicates it always applies. Total scores range from 7 to 49, with higher scores indicating greater levels of work-related psychological resilience.

SECONDARY OUTCOMES:
Physical and Physical State | Measurements will be taken before the workshop intervention, immediately after the workshop intervention, and one month later.
  We use the Single Item Fatigue Scale, scored on a Numerical Rating Scale (0-10), where 0 indicates no fatigue and 10 indicates extreme fatigue. This scale measures oncology nurses' subjective fatigue levels on the assessment day, with higher scores reflecting greater fatigue.
Physical and Physical State | Measurements will be taken before the workshop intervention, immediately after the workshop intervention, and one month later.
  We use the Depression, Anxiety, and Stress Scale - 21 Items (DASS-21) for measurement. The scale consists of 21 items, each rated on a 4-point Likert scale, where 0 indicates the symptom never applies and 3 indicates it applies most of the time or very much. Higher scores reflect greater severity of the symptoms.
Physical and Physical State | Measurements will be taken before the workshop intervention, immediately after the workshop intervention, and one month later.
  We use the Nurses' Intent to Resign Scale, which consists of 14 items rated on a 5-point Likert scale. A score of 1 indicates the statement never applies, while a score of 5 indicates it applies to a great extent. Higher scores reflect a greater intent to resign.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided